CLINICAL TRIAL: NCT06568237
Title: A Multi-centered, Double-blind, Randomized, Placebo-controlled, Parallel Group Phase 2 Study of TEV-56286 for the Treatment of Patients With Multiple System Atrophy
Brief Title: A Study to Test if TEV-56286 is Effective in Relieving Multiple System Atrophy (MSA): A Safety and Efficacy Study
Acronym: TOPAS-MSA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV56286-NDG-20039; 2023-505320-54-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple System Atrophy
Keywords: Multiple System Atrophy (MSA)
MeSH Terms: conditions — Multiple System Atrophy | interventions — 3-(1,3-benzodioxol-5-yl)-5-(3-bromophenyl)-1H-pyrazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TEV-56286 (Experimental): Orally administered capsules once daily
  Interventions: Drug: TEV-56286
- Placebo (Placebo Comparator): Orally administered capsules once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-56286 — TEV-56286 capsules administered orally
  Other Names: emrusolmin, anle138b
  Arms: TEV-56286
Drug: Placebo — Matching placebo administered orally
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of TEV-56286 administered orally for the treatment of adult participants with Multiple System Atrophy (MSA).

A secondary objective of the study is to evaluate specific efficacy parameters of TEV-56286.

Another secondary objective is to evaluate the safety and tolerability of TEV-56286.

The planned study period per participant is 56 weeks including a screening period (up to 4 weeks), a 48-week double-blind treatment period, and a follow-up visit (approximately 4 weeks after the end of the double-blind treatment period). The study duration will be approximately 27 months.

DETAILED DESCRIPTION:
We plan to open locations in the following countries: US, Israel, Italy, Spain, Germany, France, and Japan

ELIGIBILITY:
Inclusion Criteria:

* is considered to be "clinically possible" or "clinically probable" MSA as determined by the Gilman criteria
* is medically and psychiatrically stable, as indicated by medical and psychiatric history, as well as physical and neurological examination
* Females of child bearing potential (CBP) may be included only if they have a negative pregnancy test at the screening and baseline visits
* Females of CBP whose male partners are potentially fertile (ie, no vasectomy) must use highly effective birth control methods
* Males who are potentially fertile/reproductively competent (not surgically [eg, vasectomy] or congenitally sterile) and their female partners who are of CBP must use, together with their female partners, highly effective birth control methods

  * Additional criteria apply; please contact the investigator for more information

Exclusion Criteria:

* has 2 or more relatives with history of MSA, suggestive of an alternative diagnosis other than MSA
* has participated in another clinical study involving administration of an IMP within 3 months or 5 half-lives (whichever is longer) of this IMP prior to screening
* has a history of, or acknowledges, alcohol or other substance abuse in the 12 months before screening
* is a female participant who is pregnant or breastfeeding, or plans to become pregnant during the study
* has a known hypersensitivity to any components of the IMP
* is of a vulnerable population (eg, people kept in detention or jail)
* participant is using or consuming any prohibited concomitant medications within the specified exclusionary windows of this study

  * Additional criteria apply; please contact the investigator for more information

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-06-17 (Estimated)

PRIMARY OUTCOMES:
For non-EU: Change From Baseline in the Modified Unified Multiple System Atrophy Rating Scale (UMSARS) Part I Score (excluding item 11) | Baseline to Week 48
  The UMSARS is a multidimensional, validated scale for semi-quantitative clinical assessments of MSA participants. Modified UMSARS part I includes all items with the exclusion of item 11. Item scoring is scaled 0-3 using a range of 0 (no impairment) to 3 (severe impairment).
For EU: Change From Baseline in the Total UMSARS Score Part I and Part II Combined | Baseline to Week 48
  The UMSARS is comprised of 4 parts: part I, historical review of disease-related impairments, 12 items and part II, motor examination, 14 items. As UMSARS is a unified scale, each item in parts I and II achieves a single score using a range of 0 (no impairment) to 4 (severe impairment).

SECONDARY OUTCOMES:
For non-EU: Change From Baseline in the Total UMSARS Score (Part I and Part II combined) | Baseline to Week 48
For EU: Change From Baseline in the Modified UMSARS part I score (excluding item 11, item scoring rescaled 0-3) | Baseline to Week 48
Change From Baseline in the UMSARS Part 1 Score | Baseline to Week 48
Change From Baseline in Lateral Ventricle Volume Measured by MRI | Baseline to Week 48
Change From Baseline in the Clinical Global Impression - Severity scale (CGI-S) | Baseline to Week 48
  The CGI-S scale permits a global evaluation of the participant's current severity of illness on a Likert type scale ranging from 1 to 7, where 1=normal/not at all ill, 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7=among the most extremely ill participants
Change From Baseline in the Neurofilament Light Chain (NfL) Concentrations in Cerebrospinal Fluid (CSF) | Baseline to Week 48
Change From Baseline in the Patient Global Impression-Severity Scale (PGI-S) | Baseline to Week 48
  The PGI-S scale permits an evaluation of the participant's MSA severity, according to the participant. The PGI-S scale rates the participant's MSA severity on a 5-point Likert type scale ranging from 0 (not severe) to 4 (very severe)
Change From Baseline in the Pons volume measured by MRI | Baseline to Week 48
Change From Baseline in the Cerebellar volume measured by MRI | Baseline to Week 48
Change From Baseline in the UMSARS part II score | Baseline to Week 48
Change From Baseline in the UMSARS part IV score | Baseline to Week 48
Change From Baseline in the Two-minute walk test as part of gait assessment | Baseline to Week 48
Change From Baseline in the Multiple System Atrophy - Quality of Life (MSA-QoL) Score | Baseline to Week 48
  The 40-item MSA-QoL questionnaire is self-administered and each item is rated on a Likert type scale (0: No problem) to (4: Extreme problem). It is comprised of 3 subscales relevant to MSA: motor (14 items), non-motor (12 items), and emotional/social (14 items). The MSA-QoL total score is the sum of all the items and lower scores indicate better QoL.
Number of Participants With At Least One Treatment-Emergent Adverse Event (TEAEs) | Up to Week 48
Number of Participants Who Withdraw From the Study Due to an Adverse Event | Up to Week 48
Number of Participants Who Withdraw From Treatment Due to an Adverse Event | Up to Week 48
Number of Participants With At Least One Potentially Clinically Significant Abnormal Vital Sign Value | Up to Week 48
Number of Participants With At Least One Potentially Clinically Significant Laboratory Test Value | Up to Week 48
Number of Participants with at Least One Potentially Clinically Significant Change in 12-lead Electrocardiogram (ECG) Findings | Up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Tev Medical Expert, Study Director, Study Director — Teva Branded Pharmaceutical Products R&D LLC
Locations (54):
- United States (18):
  - Teva Investigational Site 15554, La Jolla, California
  - Teva Investigational Site 15545, Los Angeles, California
  - Teva Investigational Site 15547, Washington D.C., District of Columbia
  - Teva Investigational Site 15544, Boca Raton, Florida
  - Teva Investigational Site 15555, Tampa, Florida
  - Teva Investigational Site 15550, Chicago, Illinois
  - Teva Investigational Site 15546, Kansas City, Kansas
  - Teva Investigational Site 15736, Boston, Massachusetts
  - Teva Investigational Site 15870, Farmington Hills, Michigan
  - Teva Investigational Site 15552, Rochester, Minnesota
  - Teva Investigational Site 15549, New York, New York
  - Teva Investigational Site 15551, New York, New York
  - Teva Investigational Site 15553, Durham, North Carolina
  - Teva Investigational Site 15735, Hershey, Pennsylvania
  - Teva Investigational Site 15548, Pittsburgh, Pennsylvania
  - Teva Investigational Site 15869, Georgetown, Texas
  - Teva Investigational Site 15873, Alexandria, Virginia
  - Teva Investigational Site 15543, Spokane, Washington
- France (4):
  - Teva Investigational Site 35290, Bordeaux
  - Teva Investigational Site 35289, Marseille
  - Teva Investigational Site 35291, Salpêtrière
  - Teva Investigational Site 35292, Toulouse
- Germany (9):
  - Teva Investigational Site 32823, Beelitz-Heilstätten
  - Teva Investigational Site 32818, Dresden
  - Teva Investigational Site 32822, Düsseldorf
  - Teva Investigational Site 32825, Kassel
  - Teva Investigational Site 32826, Leipzig
  - Teva Investigational Site 32824, Marburg
  - Teva Investigational Site 32820, München
  - Teva Investigational Site 32819, Münster
  - Teva Investigational Site 32821, Ulm
- Israel (3):
  - Teva Investigational Site 80203, Haifa
  - Teva Investigational Site 80215, Jerusalem
  - Teva Investigational Site 80204, Tel Aviv
- Italy (6):
  - Teva Investigational Site 30299, Bologna
  - Teva Investigational Site 30297, Catania
  - Teva Investigational Site 30298, Milan
  - Teva Investigational Site 30294, Padua
  - Teva Investigational Site 30296, Roma
  - Teva Investigational Site 30295, Salerno
- Japan (7):
  - Teva Investigational Site 84140, Chiba
  - Teva Investigational Site 84139, Fuchū
  - Teva Investigational Site 84136, Gifu
  - Teva Investigational Site 84137, Niigata
  - Teva Investigational Site 84138, Sagamihara
  - Teva Investigational Site 84141, Sanda-shi
  - Teva Investigational Site 84135, Sendai
- Spain (7):
  - Teva Investigational Site 31323, Barcelona
  - Teva Investigational Site 31321, Barcelona
  - Teva Investigational Site 31324, Barcelona
  - Teva Investigational Site 31327, Madrid
  - Teva Investigational Site 31320, Pamplona
  - Teva Investigational Site 31322, Seville
  - Teva Investigational Site 31319, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

REFERENCES:
- See also: Teva MSA Trial — https://www.tevapharm.com/teva-clinical-trials/clinical-trials-results/clinical-trials/tv56286ndg20039
- See also: TOPAS-MSA Web Site — https://topas-msa-study.com/
- See also: Teva MSA Trial EU Locations — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2023-505320-54-00